CLINICAL TRIAL: NCT02945774
Title: Molecular Neuroimaging of Neuroinflammation in Neurodegenerative Dementias
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 107561
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Frontotemporal Dementia
Keywords: PET; MRI; Inflammation; Microglia; FEPPA
MeSH Terms: conditions — Frontotemporal Dementia; Inflammation | interventions — N-(2-((N-(4-phenoxypyridin-3-yl)acetamido)methyl)phenoxy)ethyl fluoride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- (18F)-FEPPA (Experimental)
  Interventions: Radiation: (18F)-FEPPA

INTERVENTIONS:
Radiation: (18F)-FEPPA — PET ligand that binds to activated microglia, a marker of neuroinflammation

SUMMARY:
Neuroinflammation is increasingly implicated as a potential critical pathogenic mechanism in a variety of neurologic and psychiatric disorders. This study will use hybrid PET/MRI imaging to evaluate neuroinflammation and its relationship to cerebral perfusion in frontotemporal dementia (FTD). Patients with FTD will be recruited from the Cognitive Neurology and Aging Brain clinics at Parkwood Institute and will undergo neurocognitive assessment and MRI/PET using the PET ligand FEPPA which binds to activated microglia, a marker of neuroinflammation. Correlations will be conducted to determine whether abnormal neuroinflammation is present in Frontotemporal dementia and whether differential patterns of neuroinflammation are present in different FTD clinical and molecular subtypes, and to determine the relationship between neuroinflammation, cerebral perfusion using arterial spin labeling MRI imaging techniques, and indices of brain structure including volumetric and white matter analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with a probable Frontotemporal Dementia or neurologically healthy control participants with no history of neurological problems
2. Study partner is available who has frequent contact with the subject and can accompany the subject to all clinic visits for the duration of the protocol.
3. Visual and auditory acuity adequate for neuropsychological testing
4. Good general health with no diseases expected to interfere with the study.
5. Subject is not pregnant, lactating, or of childbearing potential (i.e. women must be two years post-menopausal, surgically sterile or practicing an effective form of family planning
6. Willing to participate in a longitudinal imaging study at 12 months.
7. Willing to undergo MRI (3Tesla)/ PET scan (with FEPPA ligand) and no medical contraindications to MRI.

Exclusion Criteria:

1. Any significant neurologic disease other than suspected Frontotemporal Dementia that would better account for symptoms (i.e. frontal lobe stroke).
2. Screening/baseline MRI scans with evidence of infection, infarction, or other focal lesions. Subjects with multiple lacunes are excluded.
3. Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body that may preclude MRI participation as per MRI screening form.
4. Major depression, bipolar disorder as described in DSM-IV within the past 1 year. Psychotic features, agitation or behavioral problems within the last 3 months which could lead to difficulty complying with the protocol.
5. History of schizophrenia (DSM IV criteria).
6. Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol.
7. Clinically significant abnormalities in B12, or thyroid function tests that might interfere with the study.
8. Investigational agents are prohibited one month prior to entry and for the duration of the trial.
9. Exclusion for FEPPA: Current or recent participation in any procedures involving radioactive agents such that the total radiation dose exposure to the subject in any given year would exceed the limits of annual and total dose commitment set forth. The current regulation for radiation dose to patient volunteers and health control volunteers are contained within Health Canada's recently amended (June 19, 2012) Regulations Amending the Food and Drug Regulations (Positron-emitting Radiopharmaceuticals). Limitations for effective total body dose is 50 mSv (C.03.305 (c)) which has been increased from the previous values of 20 mSv (Table 1 in INFO-0491).
10. Exclusion Criteria for controls undergoing arterial line placement: Absent pulse, Thromboangiitis obliterans (Buerger disease), Burns over the cannulation site, Inadequate circulation to the extremity, Raynaud syndrome, Anticoagulation therapy, Atherosclerosis of upper extremity vessels, Coagulopathy, inadequate collateral flow, Infection at the cannulation site, Previous surgery in the area, Synthetic vascular graft.

Ages: 30 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Group differences in regional PET FEPPA ligand imaging | 120 Minutes

SECONDARY OUTCOMES:
Correlation between PET FEPPA ligand images and specified MR images | 120 Minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Parkwood Institute, London, Ontario, Canada